CLINICAL TRIAL: NCT02301845
Title: Validation of a Marker for Aspiration and Endotracheal Tube Cuff Leak.
Brief Title: Validation of Aspiration Markers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IRB disapproval
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Staff Anesthetist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Creatures
Record Dates: First submitted 2014-11-23; First posted 2014-11-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Pneumonia, Aspiration
Keywords: Respiration, artificial
MeSH Terms: conditions — Pneumonia, Aspiration; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Suspended Diatoms (Experimental): Suspended diatom shells (10 mg/ 10 ml of saline) will be instilled in the oral cavity of the study subject every 12 hours for the first three study days. The total amount of amorphous silica administered will be 20 mg/day, which is the average daily intake of amorphous silica in normal human diet (0.3 mg/kg body weight/day)
  Interventions: Drug: Diatoms Shells

INTERVENTIONS:
Drug: Diatoms Shells — Instillation of suspended diatom shells - 10 mg q12h

SUMMARY:
This is an interventional crossover study aimed at validating diatom shells as a marker for cuff leak and microaspiration in mechanically ventilated, critically ill patients.

DETAILED DESCRIPTION:
At present there is no standard method for the evaluation of in vivo cuff leak and aspiration. Most of the tested techniques have major pitfalls that render their routine application infeasible. Lacking a practical and reliable marker, any possible intervention aimed at improving cuff seal and ETT performance in order to reduce VAP occurrence is going to be hindered by the inability to truly evaluate its efficacy. Radiolabeled markers are expensive, expose the patient to considerable radiological risk, and require transport to a radiological department, which would expose critically ill patients to additional risk. Dyes have the potential to give useful information about the presence of a cuff leak, but due to persistent staining of secretions, they do not allow continuous monitoring of aspiration. Amylase detection could be a good marker of aspiration, but its ability to detect aspiration is poor even when compared to pepsin. Pepsin and bile acids have the potential to detect some of the aspirations and cuff leaks that happen daily in mechanically ventilated patients, but due to their gastrointestinal nature, they do not offer any kind of information about aspiration of contaminated oropharyngeal secretions. With this research protocol, we would like to validate the use of diatom skeletons suspended in saline as a marker for determining cuff leakage and aspiration events in an ICU population and compare its efficacy in identifying aspiration events with pepsin detection. Diatoms are a major group of algae, composing the majority of phytoplankton. Their diameter is 5-15 μm on average and 1 ml of seawater usually contains about 104 diatoms. They are unicellular organisms and their main feature is that they are enclosed within a cell wall made of amorphous silica, biopolymerized in a geometric fashion that is species-dependent. At the end of their vital cycle, diatom shells deposit at the bottom of the sea. Diatom shell deposits have been found in almost every place on Earth, and are the main component of diatomaceous earth (DE). DE is an extremely fine powder composed of diatom shells that have accumulated over thousands of years. Due to its microscopical texture and inexpensive nature, it is commonly employed as a filtering media for beverages and a drying and anti-mold agent for cereals. Diatom shells compose food-grade DE in its entirety. Due to its non-crystalline, amorphous nature, it is essentially nontoxic. Our hypothesis is that administration of 10 mg of DE suspended in 10 ml of saline into the pharyngeal cavity of intubated patients will act as a reliable marker of cuff leak and aspiration in critically ill patients. Thanks to their geometric shape, diatom shells should be easily detectable in tracheal secretions when observed under a microscope. The number of diatoms-per-field observed under a fixed magnification will allow for the detection of microaspiration in a qualitative and quantitative way. The introduction of this new, safe and inexpensive marker for evaluating ETT cuff performance and for detecting aspiration will improve the design of future studies aimed at VAP prevention

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Admission to Surgical ICUs (Ellison 4 or Blake 12);
3. Patients expected to be intubated for at least 48 hours or longer from the time of enrollment.

Exclusion Criteria:

1. High PEEP requirement at enrollment (PEEP higher than 8 cmH2O)
2. Diagnosis of ARDS (any severity)
3. Status asthmaticus
4. Current or past participation in another interventional trial conflicting with the present study;
5. Pregnant women;
6. Prisoner status;
7. Patients who had partial or total gastrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Cuff leak and microaspiration | 3 days
  The investigators will collect samples of tracheal secretions below the cuff every 4 hours after the first pharyngeal administration of diatom shells and after 12 hours from the other 5 scheduled administrations of diatom shells. Samples will be centrifuged and the sediment observed under microscopy for detection of shells in tracheal secretions below the endotracheal tube cuff. Their presence will be a sign of cuff leak and aspiration. The ratio between administered diatom shells and collected diatom shells will be used to give an estimate of leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States